CLINICAL TRIAL: NCT01032720
Title: Ultrasound-guided Versus Sham Ultrasound Corticosteroid Knee Injections
Brief Title: Ultrasound (US)-Guided Versus Sham Ultrasound Corticosteroid (CS) Knee Injections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01334
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2012-02

CONDITIONS: Osteoarthritis
Keywords: ultrasound; osteoarthritis; knee; corticosteroids; intra-articular; injections
MeSH Terms: conditions — Osteoarthritis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound-guided knee CS injection (Experimental): Ultrasound will be used to image knee joint and guide needle for intra-articular knee CS injection.
  Interventions: Procedure: Ultrasound
- Sham Ultrasound knee CS injection (Sham Comparator): CS knee injection will be performed in the same method as the US-guided knee injection but the US machine will be turned off.
  Interventions: Procedure: Sham ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound will be used to image knee joint and guide needle for intra-articular corticosteroid injection.
  Other Names: Sonosite
  Arms: Ultrasound-guided knee CS injection
Procedure: Sham ultrasound — Knee CS injection will be performed in the same method as the US-guided injection except that the US machine will be turned off. Study patient will be unaware of whether US machine is on or off.
  Other Names: Sonosite
  Arms: Sham Ultrasound knee CS injection

SUMMARY:
To determine if ultrasound-guided knee steroid injections are more effective than sham ultrasound knee steroid injections for the treatment of osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 89.
* Meet the American College of Rheumatology criteria for knee OA with knee pain, aching or stiffness on most of the past 30 days and have evidence on radiograph of a definite osteophyte.
* Have a pain score of at least 4 out of 10 on an 11 point numeric rating scale.
* For participants with bilateral knee OA, the most symptomatic knee will be considered the study knee. If both knees are symptomatic, the subject will choose the one they want treated.
* Be able to speak and understand English.
* Have a telephone.

Exclusion Criteria:

* Prior hyaluronic acid injection.
* Scheduled knee hyaluronic acid injections, arthroscopy, or knee surgery.
* Comorbid conditions including: known other causes of arthritis (infectious arthritis, rheumatoid arthritis, connective tissue disease, gout, pseudogout, or psoriatic arthritis), bony or soft tissue malignancy or skin lesions or peripheral neuropathy involving the lower extremities, cardiopulmonary disease which limits walking more than knee pain, knee instability defined as report of knee buckling or locking within the past month of the study knee, major neurologic deficit that affects gait, psychiatric illness that limits informed consent
* Current involvement in litigation or receiving workmen's compensation. These patients are to be excluded because they are expected to bias results. This group will be expected to over-report pain symptoms. This bias cannot be corrected for in the analysis.
* Contraindications to intra-articular injections: known bleeding disorder/diathesis.
* Prosthesis in the painful knee.
* Bilateral total knee replacements.
* Pregnancy if no recent knee x-rays are available.
* Wheelchair bound.
* BMI greater than 40.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Compare the effectiveness of US-guided vs. sham US CS intra-articular knee injections as measured by a 10-point between groups difference in the Knee injury and Osteoarthritis Outcome score (KOOS). | 4 weeks

SECONDARY OUTCOMES:
Compare the effectiveness of US-guided vs. sham US CS knee injections in reducing pain as measured by KOOS. | 2, 6, and 8 weeks
Compare the effectiveness of US-guided vs. sham US CS knee injections in improving self-reported lower extremity function. | 2, 4, 6, and 8 weeks
Compare the effectiveness of US-guided vs. sham US CS knee injections in reducing the proportion of patients experiencing knee pain. | 2, 4, 6, and 8 weeks
Compare the effectiveness of US-guided vs. sham US knee injections in reducing the use of co-therapies (acetaminophen, nonsteroidal anti-inflammatory drugs, and narcotics) | 2, 4, 6, and 8 weeks
Examine whether body mass index, presence or absence of chronic widespread pain, radiographic severity, patient expectations, patient satisfaction, and dispositional optimism predict response to CS injections. | 2, 4, 6, and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liana Fraenkel, M.D., Principal Investigator — VACHS; Yale University School of Medicine
Locations (1):
- West Haven Veteran's Administration Medical Center, West Haven, Connecticut, United States

REFERENCES:
- [Background] Jackson DW, Evans NA, Thomas BM. Accuracy of needle placement into the intra-articular space of the knee. J Bone Joint Surg Am. 2002 Sep;84(9):1522-7. doi: 10.2106/00004623-200209000-00003. PMID 12208907
- [Background] Hunt IM, Silman AJ, Benjamin S, McBeth J, Macfarlane GJ. The prevalence and associated features of chronic widespread pain in the community using the 'Manchester' definition of chronic widespread pain. Rheumatology (Oxford). 1999 Mar;38(3):275-9. doi: 10.1093/rheumatology/38.3.275. PMID 10325667
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Giltay EJ, Kamphuis MH, Kalmijn S, Zitman FG, Kromhout D. Dispositional optimism and the risk of cardiovascular death: the Zutphen Elderly Study. Arch Intern Med. 2006 Feb 27;166(4):431-6. doi: 10.1001/archinte.166.4.431. PMID 16505263
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558